CLINICAL TRIAL: NCT04387123
Title: Simplification of Vaginoscopic Surgery Using a Self-retaining External Vulvar Sheet (Darwish Sheet)
Acronym: Darwish sheet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Professor Atef Darwish, Prof, Woman's Health University Hospital, Egypt
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Darwish sheet
Record Dates: First submitted 2020-05-08; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Vaginoscopy
Keywords: vaginoscopy; Darwish sheet; Vagina; cervix; virgin; nullipra

STUDY DESIGN:
Intervention Model Description: Vaginoscopy via Darwish sheet or without its use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional vaginoscopy (Active Comparator): Vaginoscopy without vulvar tightness
  Interventions: Procedure: Vaginoscopy
- Tight vaginoscopy (Active Comparator): Vaginoscopy via Darwish sheet
  Interventions: Procedure: Vaginoscopy

INTERVENTIONS:
Procedure: Vaginoscopy — Vaginoscopic examination and possible operative endoscopic management

SUMMARY:
Vaginoscopic examination is usually difficult due to continuous leakage of the distension medium from the introitus. This study aims to assess the effectiveness and success of performing diagnostic or operative vaginoscopic surgery via a tight self-retaining external vulvar sheet (Darwish sheet) expressed as tight vaginoscopy (TV) compared with conventional vaginoscopy (CV).

DETAILED DESCRIPTION:
This is a prospective cross-sectional interventional cohort study was performed at the Endoscopy Unit of the Woman's Health University Hospital, Assiut, Egypt, between July 2014 and January 2020. Participants were symptomatic patients with suspected narrow vagina. They were children, adolescents or nulliparous adult females scheduled for vaginoscopy to confirm the diagnosis and whenever indicated to remove a vaginal or cervical lesion or FB. All cases underwent a high-resolution 2D transabdominal ultrasonography with full-bladder technique to assess the vaginal integrity, length and width. If a mass was seen, the examiner commented on its origin (whether cervical or vaginal), its echogenicity, and its dimensions. In doubtful cases, a pelvic MRI was requested to confirm the diagnosis. Children with suspected FB were subjected to plain X-ray to confirm the diagnosis. Patients with definite or suspected vaginal or cervical lesions were included in this study. For young girls or virgin adults, every effort was exerted to avoid hymenal injury during vaginoscopy on their request. All the cases were prepared for a vaginoscopic surgery at the regular endoscopy unit in the immediate postmenstrual period (if postmenarchal) but young girls were operated on at any time.

Every patient was subjected to a sequential diagnostic conventional vaginoscopy (CV) followed by tight vaginoscopy (TV), and whenever required operative TV. Vulvar tightness was made using a self-retaining external vulvar sheet (Darwish sheet). Under general anesthesia, all the cases were placed in the dorsal lithotomy position. Trendelenburg position was avoided because it hinders access to the entire vagina and the cervix, and may increase the risk of gas or air embolism. For adult cases, conventional hysteroscope was used as a vaginoscope. A 4-mm zero-degree telescope loaded inside a 5-mm outer sheath and connected to a light cable, with a pneumatic infusion pump for 0.9% saline irrigation, was inserted inside the vaginal introitus. At the investigator's institution, automatic infusion pumps are not used for vaginoscopic surgery as the vagina is a distensible organ unlike the uterus. The vaginoscope was gradually advanced inside the vagina (Figure 1) with reporting on the vaginal walls till the ectocervix. Proper examination of the cervix included the endocervical canal and the internal os. If feasible, the telescope was advanced to examine the endometrial cavity, searching for any associated intrauterine lesion, with a comment on the endometrial pattern and vasculature. Any suspected lesion was prepared for complete excision or at least biopsy to complete the diagnosis. On the other hand, for children, office hysteroscope (a 2.6-mm telescope and a 3.2-mm outer sheath) was used and the procedure was performed in the same way as that in adults, with exemption of uterine cavity examination. The visualized pattern of any vaginal or cervical lesion was reported. At the end of the procedure, the telescope loaded inside its sheath was extracted. The same patient was re-examined using TV. The vaginoscope penetrates a sterile self-retaining tight external silicone vulvar sheet (Darwish sheet) measuring 20x15 cm which is tied around the patient waist (Figure 2) with a central linear incision of 10 mm aiming to minimize the reflux of the irrigating fluid from the vagina. Comment on the appearance of the normal anatomy of the vagina (Figure 1) and the cervix, (Figure 3) any vaginal or cervical lesion like cervical polyps (figure 3,4) or foreign bodies (FB) (Figure 4), or a vaginal septum (video) was made. Importantly, the surgeon commented on clarity of visualization, amount of used and leaked 0.9% saline before and after application of Darwish sheet on the vulva.

For operative TV, a 27-Fr rotatory resectoscope loaded inside the sterile self-retaining tight external silicone vulvar sheet (Darwish sheet). Glycine 1.5% was used for monopolar resectoscopy. Vaginal or cervical polyps were excised by a loop electrode, while vaginal septum was cut using a hook electrode. FB was extracted using a flexible grasping forceps inserted in the vagina alongside the vaginoscope; if any difficulty was faced, the telescope was loaded inside rigid grasping forceps to extract the FB. A comment on the feasibility of surgery (clarity of visualization and access to the lesion), operative time and any possible complications was made. The amount of irrigated distension medium as well as escaped amount in the suction unit and that collected in a sterile plastic bag embedded under the buttocks of the patient were collected and measured after every case of the diagnostic CV, diagnostic TV, and operative TV. All endoscopic equipment was manufactured by Storz Co. (Tuttlingen, Germany). All excised tissues were sent for histopathologic assessment. The attached video shows different cases of diagnostic and operative vaginoscopy before and after application of Darwish sheet. The main outcome measures included clarity of visualization of the vagina and the cervix, estimation of infused and leaked distension medium before and after application of vulvar Darwish sheet and the success rate of operative TV whenever indicated. Postoperatively, the patients were kept under observation for 2-4 h and discharged whenever stable. All cases were followed up at least once after the next menses and examined clinically and by ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

children, adolescents nulliparous adult females scheduled for vaginoscopy Suspected vaginal or cervical lesion or foreign body FB

Exclusion Criteria:

Multiparous patients nulliparous patients with normal, patulous or lax vaginas

Ages: 4 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
clarity of visualization of the vagina and the cervix | 1 day
  clear
estimation of infused and leaked distension medium before and after application of vulvar Darwish sheet | 1 day
the success rate of operative TV whenever indicated | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Woman's Health University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No